CLINICAL TRIAL: NCT01442181
Title: Minimally Invasive Surgical Treatment Versus Medical Management for Stroke Patients With Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 433-2009; NCT01413971 (obsolete NCT alias)
Record Dates: First submitted 2010-10-05; First posted 2011-09-28 (Estimated); Results first posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Atrial Fibrillation; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Minimally Invasive Surgical Procedures; Nutrition Therapy; Practice Management, Medical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minimally Invasive Surgery (Active Comparator): Thumb sized incisions are made on each sides of the chest wall where instruments are placed in the chest to perform the surgery.
  Interventions: Procedure: Minimally Invasive Surgery
- Medical Therapy (Active Comparator): Patients are treated with rhythm and rate control medications.
  Interventions: Other: Medical therapy

INTERVENTIONS:
Procedure: Minimally Invasive Surgery — Small thumb sized incisions are made on each side of the chest wall where instruments are inserted for the purpose of completing the surgery.
  Other Names: Minimally Invasive Maze Procedure
  Arms: Minimally Invasive Surgery
Other: Medical therapy — Patients are treated with rhythm and rate control medications.
  Other Names: Medical Management
  Arms: Medical Therapy

SUMMARY:
The purpose of this study is to compare a minimally invasive surgical procedure and medication management in stroke patients with Atrial Fibrillation. The two treatment options are a minimally invasive surgical procedure or the use of medications.

DETAILED DESCRIPTION:
Must have had a stroke or transient ischemic attack (TIA) and have Atrial Fibrillation

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of stroke and paroxysmal, persistent or permanent AF.
* Ischemic stroke or TIA with documented paroxysmal or persistent atrial fibrillation. A TIA will meet inclusion criteria as a sudden-onset focal neurological symptom or sign lasting at least 10 minutes but less than 24 hours with or without evidence of acute brain ischemia on diffusion weighted MRI imaging.
* Eligible symptoms INCLUDE hemiplegia or hemiparesis, monoplegia, or language disturbance other than isolated dysarthria.
* Symptoms that will NOT QUALIFY AS TIA INCLUDE transient monocular blindness in both eyes, dysarthria, vertigo,isolated sensory symptoms, confusion, memory loss, nonspecific complaints of dizziness, or syncope.

Exclusion Criteria:

* Recent stroke (< 1 month).
* Age < 18 or > 80 years; Ejection Fraction < 25%• Presence of left atrial appendage thrombus on CT or echocardiography
* Previous empyema or thoracic surgery, preventing access to the pulmonary veins via thoracoscopy.
* Left Atrial Diameter > 55mm.
* Contraindication to anticoagulation with Coumadin.
* Mitral insufficiency (> 2+)
* • • Contraindications to MRI
* •Artificial heart valve prosthesis
* Aneurysm clips
* Implanted drug infusion device or pump
* Any type of neurotranstimulator
* Any type of bone growth stimulator
* Cochlear implants or inner ear prosthesis
* Any intravascular coils, filters, or stents
* Shrapnel or bullets
* Other metallic implants or devices specify which
* Permanently tattooed eyeliner
* Are you pregnant or suspect to be pregnant?

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-03; Primary Completion 2013-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Beaver, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Minimally Invasive Surgery | Medical Therapy
Started | 14 | 11
Completed | 10 | 8
Not Completed | 4 | 3
Not completed — patient refused surgery | 1 | 0
Not completed — no insurance for surgery | 1 | 0
Not completed — low ejection factor | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — patient in an additional study | 1 | 0
Not completed — atrial fibrillation not noted | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minimally Invasive Surgery | Medical Therapy | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 9 | 8 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  United States | 14 | 11 | 25

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life RAND 36-Item Health Survey
Description: Compare quality of life of patient satisfaction between the surgery and or the medication in stroke patients with AF (atrial fibrillation).
  The RAND 36-Item Health Survey taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. Note that all items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. Items in the same scale are averaged together to create the 8 scale scores which will have a 0 to 100 range.
Time Frame: Change in baseline, 3 month, and 6 month
Population: Patients with ischemic stroke or transient ischemic attack (TIA) with documented paroxysmal or persistent atrial fibrillation were eligible for the study if they demonstrated the following symptoms: hemiplegia or hemiparesis, monoplegia, or language disturbance.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Minimally Invasive Surgery | Medical Therapy
Number analyzed (Participants) | 10 | 8
units on a scale
  Baseline-Energy/fatigue | 33 (19.8) | 46.25 (25.4)
  3month-Energy/fatigue | 49.5 (20.6) | 49.16 (23.1)
  6month-Energy/fatigue | 55.5 (14.4) | 54.37 (22.1)
Statistical Analysis 1: Comparison: Minimally Invasive Surgery; Energy and fatigue 3 month vs 6 month in minimally invasive group; Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Minimally Invasive Surgery; Comparison of the fatigue and energy was done in baseline-3 month, and 6 month in each group. Minimally Invasive: baseline vs 3 month; Test type: Superiority or Other; p = 0.01, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Medical Therapy; Energy and fatigue in medical therapy group; baseline vs 3 month; Test type: Superiority or Other; p = 0.49, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Medical Therapy; Energy and fatigue 3 month vs 6 month; Test type: Superiority or Other; p = 0.06, Wilcoxon (Mann-Whitney)

2. Other Pre Specified Outcome: STAI-FormY-1 Questionnaire (State-Trait Anxiety Inventory)
Description: Compare quality of life of patient satisfaction between the surgery and or the medication in stroke patients with AF (atrial fibrillation). Scores range from 20 to 80, with higher scores correlating with greater anxiety.
Time Frame: Change in baseline, 3 month, and 6 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Minimally Invasive Surgery | Medical Therapy
Number analyzed (Participants) | 10 | 8
units on a scale
  Baseline | 41.20 (9.76) | 37.5 (8.68)
  3 month | 35.7 (10.88) | 35.00 (14.05)
  6 month | 35.67 (11.54) | 42.38 (9.86)

3. Other Pre Specified Outcome: STAI-Form-Y2 Questionnaire (State-Trait Anxiety Inventory)
Description: as for outcome 2
Time Frame: Change in baseline, 3 month, and 6 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Minimally Invasive Surgery | Medical Therapy
Number analyzed (Participants) | 10 | 8
units on a scale
  Baseline | 38.20 (10.50) | 40.50 (10.77)
  3 month | 36.50 (11.65) | 34.88 (12.64)
  6 month | 35.00 (10.69) | 35.38 (8.40)

4. Other Pre Specified Outcome: Montreal Cognitive Assessment (Moca)
Description: Compare quality of life of patient satisfaction between the surgery and or the medication in stroke patients with AF (atrial fibrillation). The score is 0 - 30 point test with the higher the score the better cognitive function.
Time Frame: Change in baseline, 3 month, and 6 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Minimally Invasive Surgery | Medical Therapy
Number analyzed (Participants) | 10 | 8
units on a scale
  Baseline | 25.89 (3.55) | 23.25 (6.92)
  3 month | 26.44 (2.35) | 24.86 (5.93)
  6 month | 25.33 (4.36) | 24.38 (5.73)

5. Other Pre Specified Outcome: Directed Fluency; Cowa (Controlled Oral Word Association Test)
Description: Compare quality of life of patient satisfaction between the surgery and or the medication in stroke patients with AF (atrial fibrillation). The participant is asked to name as many words as possible beginning with a letter, excluding proper nouns, for one minute and this procedure is repeated three times.
Time Frame: Change in baseline, 3 month, and 6 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Minimally Invasive Surgery | Medical Therapy
Number analyzed (Participants) | 10 | 8
words
  COWA, baseline | 39.70 (9.23) | 29.38 (14.34)
  COWA, 3 month | 44.33 (12.12) | 27.00 (11.12)
  COWA, 6 month | 41.40 (10.30) | 28.25 (11.27)

6. Other Pre Specified Outcome: Hopkins Verbal Learning Test Version A
Description: Compare quality of life of patient satisfaction between the surgery and or the medication in stroke patients with AF (atrial fibrillation). This test measures word recognition. 12 words are read to the subject and they have to repeat as many as they can recall. There are 4 trials, each with 12 total possible words.
Time Frame: Change in baseline, 3 month, and 6 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Minimally Invasive Surgery | Medical Therapy
Number analyzed (Participants) | 10 | 8
words
  HVLT 1_baseline | 4.70 (2.06) | 4.38 (1.41)
  HVLT 1_3 month | 6.00 (1.41) | 4.14 (1.77)
  HVLT 1_6 month | 6.00 (2.55) | 4.13 (2.42)
  HVLT 2_baseline | 5.50 (2.80) | 5.88 (1.96)
  HVLT 2_3 month | 7.67 (2.50) | 5.14 (2.85)
  HVLT 2_6 month | 6.44 (3.00) | 5.75 (2.71)
  HVLT 3_baseline | 7.10 (3.00) | 6.13 (3.14)
  HVLT 3_3 month | 7.44 (3.40) | 6.29 (2.14)
  HVLT 3_6 month | 6.78 (2.99) | 6.63 (1.85)
  HVLT Total_baseline | 17.30 (7.02) | 16.38 (5.93)
  HVLT Total_3 month | 21.11 (6.94) | 15.57 (6.08)
  HVLT Total_6 month | 19.22 (8.21) | 16.50 (6.72)

7. Other Pre Specified Outcome: Stroop Color Test
Description: Compare quality of life of patient satisfaction between the surgery and or the medication in stroke patients with AF (atrial fibrillation). Only 9 patients in the minimally invasive surgery arm completed the stroop color test, and only 6 patients in the medical therapy group completed the stroop color test.
  In this test, subjects are asked to read a list of color words. 100 is the maximum amount of correct responses per trial.
Time Frame: Change in baseline, 3 month, and 6 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: colors
Arm/Group | Minimally Invasive Surgery | Medical Therapy
Number analyzed (Participants) | 9 | 6
colors
  Stroop color_baseline | 57.89 (13.32) | 53.33 (8.36)
  Stroop color_3 month | 58.14 (16.41) | 53.50 (4.51)
  Stroop color_6 month | 50.00 (9.06) | 47.60 (19.11)

8. Other Pre Specified Outcome: Wtar (Wechsler Test of Adult Reading) Word List
Description: Compare quality of life of patient satisfaction between the surgery and or the medication in stroke patients with AF (atrial fibrillation).
  The WTAR is composed of 50 irregularly spelled words and takes approximately 10 minutes to complete. The examiner begins by presenting the first word card and prompting the patient for a single pronunciation of the word. This procedure continues through all 50 word cards and is discontinued if the patient provides 12 consecutive incorrect pronunciations. Each correct pronunciation is given a score of 1, with 50 as the maximum raw score.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Minimally Invasive Surgery | Medical Therapy
Number analyzed (Participants) | 10 | 8
words | 40.50 (9.40) | 32.50 (7.75)

9. Other Pre Specified Outcome: Stroop Word Test
Description: Compare quality of life of patient satisfaction between the surgery and or the medication in stroke patients with AF (atrial fibrillation). Only 9 patients in the minimally invasive surgery arm completed the stroop word test, and only 6 patients in the medical therapy group completed the stroop word test.
  In this test, subjects are asked to read a list of words. 100 is the maximum amount of correct responses per trial.
Time Frame: Change in Baseline, 3 month, and 6 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Minimally Invasive Surgery | Medical Therapy
Number analyzed (Participants) | 9 | 6
words
  Stroop word_Baseline | 74.78 (16.74) | 75.33 (15.32)
  Stroop word_3 month | 80.71 (12.16) | 75.75 (7.27)
  Stroop word_6 month | 76.00 (8.00) | 66.60 (24.14)

10. Other Pre Specified Outcome: Directed Fluency, Animals
Description: Compare quality of life of patient satisfaction between the surgery and or the medication in stroke patients with AF (atrial fibrillation). The participant is asked to name as many animals as possible beginning with a letter, for one minute.
Time Frame: Change in Baseline, 3 month, and 6 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: animals
Arm/Group | Minimally Invasive Surgery | Medical Therapy
Number analyzed (Participants) | 10 | 8
animals
  Animals, baseline | 18.10 (6.35) | 15.75 (5.65)
  Animals, 3 month | 17.89 (4.20) | 15.00 (5.23)
  Animals, 6 month | 17.70 (7.24) | 14.50 (5.68)

ADVERSE EVENTS:
Time Frame: For the duration of treatment, up to 6 months
Arm/Group | Minimally Invasive Surgery | Medical Therapy
Serious Adverse Events (participants affected / at risk) | 2/14 | 0/11
Other Adverse Events (participants affected / at risk) | 6/14 | 2/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minimally Invasive Surgery (N=14) | Medical Therapy (N=11)
thrombus left appendage (Cardiac disorders) | 1 (1) | 0 (0) — case was canceled on the OR table due to clot in left appendage
extensive pericardial adhesions (Cardiac disorders) | 1 (1) | 0 (0) — case was canceled due to extensive pericardial adhesions
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minimally Invasive Surgery (N=14) | Medical Therapy (N=11)
imbalance and moemory loss (Nervous system disorders) | 1 (1) | 1 (1) — Head MRI and head CT were done both normal
passed out (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — passed out at home was transported to ER was diagnosed with dehydration
external cardioversion (Cardiac disorders) | 3 (3) | 0 (0) — atrial fibrillation
open wound (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) — open wound incision sites, home health care with wet to dry packing
tachycardia (Cardiac disorders) | 1 (1) | 0 (0) — fast heart rate, medication change and patient monitored

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No